CLINICAL TRIAL: NCT04862260
Title: A Phase 1 Feasibility Study of Cholesterol Metabolism Reprogramming (Evolocumab, Atorvastatin and Ezetimibe) in Combination With the Standard of Care in Patients With Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Cholesterol Disruption in Combination With the Standard of Care in Patients With Advanced Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Biovalorem (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLOE pancreas
Record Dates: First submitted 2021-04-06; First posted 2021-04-27 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Pancreas Cancer; Metastatic Cancer
Keywords: Statin; Atorvastatin; Lipitor; PCSK9 monoclonal antibody; PCSK9 inhibitor; PCSK9; Evolocumab; Repatha; Alirocumab; Praluent; Lipid droplets and vacuoles; NPC1L1 transporter; HMG Co A reductase; LDL receptor; LRP1 receptor; SRB1 receptor; Lipids; Cancer; Cholesterol; Pancreas cancer; Pancreas/Pancreatic Cancer Metastatics; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Hyperlipoproteinemia Type II; Neoplasms | interventions — Atorvastatin; Ezetimibe; evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Multipathway cholesterol metabolism disruption (Experimental): Twelve to fifteen patients will receive a combination of daily atorvastatin 40 mg, twice daily ezetimibe 10 mg and evolocumab 420 mg subcutaneously every month. This multipathway cholesterol metabolism disruption will be combined to standard chemotherapy (FOLFIRINOX).
  Interventions: Drug: Cholesterol metabolism disruption

INTERVENTIONS:
Drug: Cholesterol metabolism disruption — Cholesterol metabolism disruption using a combination of atorvastatin, ezetimibe and evolocumab in metastatic pancreatic adenocarcinomas
  Other Names: A combination of a lipophilic statin (Atorvastatin, Lipitor), a NPC1L1 inhibitor (Ezetimibe, Ezetrol) and a PCSK9 inhibitor (Evolocumab, Repatha) with chemotherapy in pancreatic cancer

SUMMARY:
Cardiovascular diseases and cancers, the two leading causes of death in Canada, require cholesterol to sustain their progression. All cells require cholesterol, but cancer cells have much higher needs to sustain growth, division and metastasis. The availability of new cholesterol-lowering drugs developed to protect patients from heart diseases has resulted in unprecedented low levels of cholesterol. The combination of atorvastatin, ezetimibe and Repatha, which are 3 cholesterol-lowering drugs used in combination, is safe, well tolerated and efficient over years of treatment. Recent reports indicate that abundant cholesterol supplies are required to sustain the progression of pancreatic ductal adenocarcinomas. This proof-of-concept study aims to verify the feasibility, the acceptability and gain preliminary data on adding a cholesterol shortage on top of FOLFIRINOX (standard chemotherapy) in newly diagnosed patients with locally advanced pancreatic adenocarcinomas or metastatic pancreatic adenocarcinomas. It is expected that a drug-induced cholesterol shortage will slow-down or stop the progression of pancreatic adenocarcinomas while increasing the response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to this trial, patients must fulfill the following inclusion criteria:

1. Have a histologically confirmed, treatment-naive locally advanced and inoperable (LaiPDAC) or metastatic pancreatic ductal adenocarcinoma (mPDAC).
2. Be at least 18 years or older at the time of signing the informed consent.
3. Have a life expectancy of at least 12 weeks.
4. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
5. Have measurable disease as assessed by RECIST v1.1.
6. Agrees and amenable to a tumor (if deemed safe only) and liver biopsy (all participants) at baseline and on day 42 +/- 3 days. Patient that are anticoagulated at baseline are eligible provided it is deemed safe by the investigator to stop anticoagulation momentarily in order to safely proceed to a biopsy.
7. Eligible to standard-dose FOLFIRINOX as assessed by the principal investigator or a sub-investigator. FOLFIRINOX doses can be adapted according to SOC.
8. Demonstrate normal organ function as defined below. These assessments must be done within 7 days of Cycle 1 Day-7.

   Hemoglobin (Hb) ≥ 90 g/L Absolute neutrophil count ≥ 1.5 x 10 9/L Platelet count ≥ 100 x 10 9/L INR ≤ 1.3 (unless patient is anticoagulated*) aPTT ≤ 1.5 x ULN (switching to LMWH will be recommended) Total bilirubin ≤ 1.5 x ULN OR Direct bilirubin (for patients with total bilirubin ≥ 1.5 x ULN) AST and ALT ≤ 3 x ULN CPK ≤ 1.5 x ULN Serum creatinine ≤ 1.5 x ULN OR Estimated GFR (as per institutional standards) ≥ 50 ml/min
9. Provide written informed consent and able to follow the trial treatment and visit schedule.
10. For Women Of Child-Bearing Potential (WOCBP), a negative serum pregnancy test must be obtained prior to receiving the study medication.
11. WOCBP should agree to use 2 different methods of birth control OR abstain from heterosexual intercourse for the duration of the trial and up to 90 days after the last study medication administration.
12. Male subjects should agree to use an adequate method of contraception for the duration of the trial and up to 90 days after the last study medication administration. Male subjects should refrain from donating sperm during this period.

Exclusion Criteria:

To be eligible to this trial, patients must not fulfill any of the following exclusion criteria:

1. Locally advanced pancreatic ductal adenocarcinoma deemed operable.
2. Any pancreatic ductal adenocarcinoma deemed operable or borderline operable that can be treated with neoadjuvant chemotherapy.
3. Known additional malignancy that is progressing or that requires treatment. Exceptions include basal cell carcinoma of the skin, in situ bladder or in situ cervical cancer. Other malignancy may be eligible after consultation with the promotor-investigator.
4. Spinal cord compression or brain metastases unless treated, stable and not requiring steroids for at least 4 weeks prior to the initiation of study treatment.
5. Baseline myalgia or myositis of any etiology.
6. Prior treatment with FOLFIRINOX in the adjuvant setting.
7. History of clinically significant intolerance or myositis with any statin.
8. History of clinically significant intolerance or hypersensitivity to PCSK9 inhibitors or ezetimibe.
9. Baseline grade ≥ 2 ULN Creatine Phosphokinase (CPK) elevation.
10. Liver tumor burden that is deemed unsafe by the investigator.
11. Major surgery or procedure from which the patient has not yet recovered.
12. Any medical condition that puts the patient at high medical risk, including but not limited to active uncontrolled infection or active bleeding diathesis.
13. Any history of disease that, in the opinion of the investigator, puts liver function at risk including but not limited to autoimmune hepatitis or history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Screening at baseline for those conditions is not required.
14. Use of any drugs that are contraindicated as per protocol and that cannot be changed or modified to an acceptable alternative.
15. Active smoker. Complete usage of tobacco must have been stopped for at least 3 months.
16. Abnormally low hematocrit, as assessed by the oncologist.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the rate of adverse events | 2 years
  To determine causality and grading severity of each adverse event (AEs) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Characterization of dose-limiting toxicities | 2 years
  To determine the dose at which no more than 1 out of 6 patients experience a drug related dose-limiting toxicity. To confirm that the combination of daily atorvastatin 40 mg, ezetimibe 10 mg twice daily and monthly evolocumab 420 mg meets the criterion to be the recommended phase II dose (RP2D).

SECONDARY OUTCOMES:
LDLR (low-density lipoprotein receptor) tumoral and hepatic changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of LDLR in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.
LRP1 (Low-density lipoprotein Receptor-Related Protein 1) tumoral and hepatic changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of LRP1 in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.
NPC1L1 (Niemann-Pick C1-Like 1 protein) tumoral and hepatic changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of NPC1L1 in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.
SRB1 (Scavenger Receptor class B type 1) tumoral and hepatic changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of SRB1 in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.
MHC-1 (Major Histocompatibility Complex class 1) tumoral and hepatic changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of MHC-1 in the tumor (hepatic metastasis ) and the liver by immunohistochemistry
PD-L1 (Programmed Death-Ligand-1) changes in response to the multipathway cholesterol embargo. | 1 year
  Assessment of the level of PD-L1 (Programmed Death-Ligand-1) in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.
Change in tumoral and hepatic levels of TILs (Tumor-Infiltrating Lymphocytes) | 1 year
  Assessment of tumoral and hepatic levels of TILs by immunohistochemistry
CD36 (Cluster of Differentiation 36) changes in response to the multipathway cholesterol embargo | 1 year
  Assessment of tumoral and hepatic levels in the tumor (hepatic metastasis ) and the liver by immunohistochemistry.

OTHER OUTCOMES:
Investigation of changes in the lipid profile induced by the addition of cholesterol-lowering drugs to FOLFIRINOX in metastatic pancreatic ductal adenocarcinomas (mPDAC) patients. | 1 year
  Changes in Total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides using serial assessment. All measures are in mmol/L.
Investigation of changes in circulating apo B levels induced by the addition of cholesterol-lowering drugs to FOLFIRINOX in locally advanced or metastatic pancreatic ductal adenocarcinomas (mPDAC) patients. | 1 year
  Changes in Apolipoprotein B (g/L) using serial assessment.
Investigation of changes in Apo A1 levels induced by the addition of cholesterol-lowering drugs to FOLFIRINOX in locally advanced or metastatic pancreatic ductal adenocarcinomas (mPDAC) patients. | 1 year
  Changes in Apolipoprotein A1 (g/L) using serial assessment.
Investigation of changes in PCSK9 induced by the addition of cholesterol-lowering drugs to FOLFIRINOX in locally advanced or metastatic pancreatic ductal adenocarcinomas (mPDAC) patients. | 1 year
  Changes in total, free and phosphorylated PCSK9 (Proprotein Convertase Subtilisin/Kexin type 9, ng/L) levels using serial assessment (measured by mass spectrometry).
Efficacy as measured by objective response rate | 1 year
  To obtain a preliminary assessment of the efficacy of the combination of cholesterol metabolism disruption and FOLFIRINOX: tumoral response assessment will be centrally Evaluated using RECIST v1.1.
Efficacy as measured by overall survival | 1 year
  Overall Survival (OS) at 1 year
Efficacy as measured by progression free survival | 1 year
  Progression Free Survival (PFS) at 1 year
Investigation of changes in insulin, phytosterols, ANGPTL3, ANGPTL4, ANGPTL8 and Apo C3 levels induced by the addition of cholesterol-lowering drugs to FOLFIRINOX in locally advanced or metastatic pancreatic ductal adenocarcinomas (mPDAC) patients. | 1 year
  Changes in insulin, phytosterols, ANGPTL3, ANGPTL4, ANGPTL8 and Apo C3 levels
To explore the feasibility of a larger multicenter trial | 1 year
  Collect preliminary data permitting to obtain estimates for the feasibility of a larger multicenter trial :
  Recruitment time Retention and dropout rates Acceptability of the regimen as assessed by patients Dose-limiting toxicities Response of biomarkers RECIST assessment Estimates for overall response rate (ORR) Estimates of progression-free survival (PFS) at 1 year Estimates of median overall survival (mOS) Monitor adverse effects Identification of missing data Identification of barriers to study completion Estimates to guide samples size / power calculation for a larger multicenter trial

CONTACTS AND LOCATIONS:
Overall Officials: Anne Gangloff, MD PhD FRCPC, Study Chair — CHU de Québec-Université Laval; Maxime Chénard-Poirier, MD FRCPC, Principal Investigator — CHU de Québec-Université Laval; Félix Couture, MD FRCPC, Study Director — CHU de Québec-Université Laval; Vincent Castonguay, MD FRCPC, Study Director — CHU de Québec-Université Laval; Olivier Dumas, MD FRCPC, Study Director — CHU de Québec-Université Laval; Anne-Marie Carreau, MD FRCPC, Study Director — CHU de Québec-Université Laval; Frédéric Calon, PhD, Study Director — CHU de Québec-Université Laval; Nabil G. Seidah, PhD, Study Director — Institut de recherches cliniques de Montréal; Francine Aubin, MD FRCPC, Principal Investigator — CHUM
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided